CLINICAL TRIAL: NCT06759675
Title: Comparative Effects of Group Based Exercises with and Without Cognitive Functional Therapy on Clinical Outcomes in Patients with Chronic Low Back Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Faisalabad (Other)
Responsible Party: Principal Investigator, Kashaf Zahra, Comparative effects of Group based exercises with and without Cognitive Functional Therapy on clinical outcomes in patients with chronic Low Back Pain, University of Faisalabad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GBE and CFT in chronic LBP
Record Dates: First submitted 2024-12-28; First posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-12

CONDITIONS: Low Back Pain, Chronic
Keywords: Cognitive Functional therapy; group based exercise; chronic low back
MeSH Terms: conditions — Low Back Pain; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Experimental): group based exercises with Cognitive functional therapy
  Interventions: Other: group based exercise with Cognitive functional therapy
- Group 2 (Active Comparator): group based exercise only
  Interventions: Other: Group based exercise

INTERVENTIONS:
Other: group based exercise with Cognitive functional therapy — 1. Cognitive functional therapy CFT A cognitive functional therapy is the behavioral approach which is used to treat low back pain. This approach has 3 components Making sense of pain Exposure with control Lifestyle changes
  2. Group exercises Group exercises will be the exercises that perform on all individuals. It is performed in a group session having 3 components Pain education Exercises Relaxation
  Arms: Group 1
Other: Group based exercise — Group exercises Group exercises will be the exercises that perform on all individuals. It is performed in a group session having 3 components Pain education Exercises Relaxation
  Arms: Group 2

SUMMARY:
1.1Research objective The objective of the study is to find the comparative effects of group based exercises with and without cognitive functional therapy on clinical outcomes in patients with chronic low back? 1.2 Hypothesis Null Hypothesis H0= There is no significant difference of clinical outcomes between the cognitive functional therapy with group exercises and group based exercises only in patients with chronic low back pain.

Alternative Hypothesis H1= There is a significant difference of clinical outcomes between the cognitive functional therapy with group exercises and group based exercises only in patients with chronic low back pain.

DETAILED DESCRIPTION:
Background: Low back pain is the problem gradually increasing in both young and older adults. It can be specific and non-specific, the specific low back pain is the pain which arises due to any structural or functional disease like due to any mechanical factors, poor posture, improper way of lifting and bending while non-specific low back pain is the pain which have no any known causes. Cognitive functional therapy and group based exercises both have beneficial effects to reduce LBP. Aims and objectives: The aim of the study will be to find the comparative effects of group based exercises with and without cognitive functional therapy on clinical outcome in patients with chronic low back pain. Methodology: This study will be Randomized controlled trial. The subjects will be selected through Probability Purposive Sampling.Sample will be 40 calculated by the rao-soft with 20 percent chances of drop out. The participants will be taken from Mujahid hospital, Faisal Hospital and Madina teaching hospital. Participants will be assessed by using Oswestry Disability index and Numerical Pain Rating Scale NPRS for low back pain. Participants will be randomly allocated into two groups.One group will be treated with CFT and group based exercises and one with only group exercises. And at the end, data will be analyzed by using Statistical Package for the Social Sciences (SPSS).

ELIGIBILITY:
Inclusion Criteria:

* Pain level equal or more than 3 on NPRS A score of fourteen percent 14% or more on the Oswestry Disability Index (ODI) Low back pain for at least 6months duration

Exclusion Criteria:

* Red flags (neoplastic diseases or cancer in the spine, inflammatory diseases, infections, and fractures) Neurological symptoms and psychiatric, rheumatologic, and cardiac diseases Radiculopathy with symptoms Lumbar stenosis Spondylolisthesis History of spinal surgeries Pregnancy

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
NPRS | Baseline
  Numerical pain rating scale used to assess pain level

SECONDARY OUTCOMES:
ODI | Baseline
  Oswestry Disability Index gives information about functional limitation and level of disability due to pain

IPD SHARING:
Plan to Share IPD: No
Because every participants don't want to share and this will be written in the informed consent that their data will not shared

REFERENCES:
- [Background] Oiestad BE. Critically appraised paper: Cognitive functional therapy reduced disability compared with group-based exercise and education for chronic low back pain [synopsis]. J Physiother. 2021 Apr;67(2):141. doi: 10.1016/j.jphys.2021.01.004. Epub 2021 Mar 17. No abstract available. PMID 33744183
- [Background] Avila L, da Silva MD, Neves ML, Abreu AR, Fiuza CR, Fukusawa L, de Sa Ferreira A, Meziat-Filho N. Effectiveness of Cognitive Functional Therapy Versus Core Exercises and Manual Therapy in Patients With Chronic Low Back Pain After Spinal Surgery: Randomized Controlled Trial. Phys Ther. 2024 Jan 1;104(1):pzad105. doi: 10.1093/ptj/pzad105. PMID 37548608
- [Background] O'Keeffe M, O'Sullivan P, Purtill H, Bargary N, O'Sullivan K. Cognitive functional therapy compared with a group-based exercise and education intervention for chronic low back pain: a multicentre randomised controlled trial (RCT). Br J Sports Med. 2020 Jul;54(13):782-789. doi: 10.1136/bjsports-2019-100780. Epub 2019 Oct 19. PMID 31630089